CLINICAL TRIAL: NCT05025007
Title: The Evaluation of Medial Longitudinal Arch Morphology in Children With Spastic Diplegic Cerebral Palsy by Arch Height Index Measurement Method: A Pilot Study
Brief Title: The Evaluation of Medial Longitudinal Arch Morphology in Children With Spastic Diplegic Cerebral Palsy by Arch Height Index Measurement Method
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Levent Karataş, Medical Doctor, Principal Investigator, Gazi University
Other Study IDs: Cerebral Palys and Foot
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Diplegic Cerebral Palsy With Spasticity; Pes; Deformity
Keywords: Cerebral Palys; Children; Arch Height Index; Medial Longitudinal Arch; Pes Planus; Pes Cavus; Flatfoot; Foot Deformity
MeSH Terms: conditions — Foot Deformities, Congenital; Flatfoot; Talipes Cavus; Foot Deformities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: The study cohort will consist of patients with spastic diplegic cerebral palsy who were admitted to our outpatient and inpatient clinics of the Physical Medicine and Rehabilitation Department.

SUMMARY:
Foot deformities are one of the most common orthopedic problems in patients with cerebral palsy(CP). Various methods have been proposed to evaluate foot morphology. Arch height index (AHI) measurement is a simple and quantitative method that can be applied in outpatient settings to evaluate the morphology of the medial longitudinal arch(MLA) of the foot. In this study, we aim to investigate the feasibility of AHI measurement in children with CP and, to identify other clinical findings that may be related to foot arch height determined by the AHI method.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a posture, movement, and motor dysfunction that occurs as a result of non-progressive damage of the developing brain during the intrauterine period or early childhood. Foot deformities, including pes planus and pes cavus, are common in children with CP and deteriorate posture and mobility due to its progressive nature and accompanying pain. Spasticity, muscle imbalances, soft tissue changes, and subsequent skeletal disorders are blamed for foot deformities in patients with CP.

Some methods such as foot posture index, navicular drop test, footprint methods, and radiological imaging have been described to identify and evaluate the MLA and foot/ankle posture. Arch height index (AHI) measurement is a novel method that evaluates especially medial longitudinal arch(MLA) morphology, with proven validity and reliability. It is essentially based on the measurement of the dorsum height and the length of the foot by using various caliper systems during varying degrees of load-bearing like sitting or standing. AHI measurement has some advantages over other methods. Measuring AHI during varying degrees of load-bearing such as sitting or standing allows us to quantitatively assess the mobility of the MLA. AHI measurement should be preferred in patients with foot sole skin disorders where footprint measurement methods are inefficient. Its results are not affected by some factors such as x-ray tube angle differences in foot radiography. It does not pose a risk of radiation exposure and is easy to apply. However, there is no data on the effectiveness of the AHI method in determining the MLA morphology in children with CP.

The first hypothesis of this study is that AHI measurement results in patients with CP correlate with data obtained from standard foot radiographs. The second aim of the study is to investigate the relationship between MLA morphology and other findings such as joint range of motion and spasticity of lower extremity muscles in patients with CP.

Patients with spastic diplegic cerebral palsy who were admitted to the Physical Medicine and Rehabilitation Department of our hospital will be evaluated in terms of eligibility criteria for the study. Eligible patients will be informed about the trial, and informed consent will be obtained from those who agree to participate. It was planned to recruit 24 subjects with a correlation coefficient of 0.8, a power of 0.90, and a margin of error of 0.05 to determine the correlation between AHI and quantitative foot radiography data.

Demographic data, body mass indexes, physical examination findings including gait patterns, ankle and foot range of motion and tone of the certain lower extremity muscles of participants will be recorded. MLA morphology will be evaluated by foot radiographs and AHI measurements. The AHI measurement will be made both in the bipedal standing and in the sitting position with both feet calmly on the ground. AHI will be calculated by proportioning the height of the dorsum measured from the middle 1/2 of the total length of the foot to truncated foot length.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with spastic diplegic cerebral palsy
* Being between the ages of 5-17
* Agree to participate in the study

Exclusion Criteria:

* Excessive spasticity and Achilles contracture that prevents heel contact during stance
* Botulinum toxin injection into the calf muscles in the last 3 months
* Prior orthopedic surgery of the Achilles tendon, foot, or ankle
* Radiculopathy, plexus, or peripheral nerve disorder involving the lower extremities

Ages: 60 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study cohort will consist of patients with spastic diplegic cerebral palsy who were admitted to our outpatient and inpatient clinics of the Physical Medicine and Rehabilitation Department. Every subject meeting the criteria of inclusion is going to be included in the study via a consecutive participant sampling method.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Arch Height Index while bipedeal standing | Initial evaluation of the participant
  The ratio of the height of the dorsum measured from the middle 1/2 of the total length of the foot to truncated foot length while bipedal standing
Arch Height Index while sitting | Initial evaluation of the participant
  he ratio of the height of the dorsum measured from the middle 1/2 of the total length of the foot to truncated foot length while sitting with feet calmly on the ground
Navicular Index | Initial evaluation of the participant
  The ratio of the height of the navicular bone from the ground to the height of the medial longitudinal arch of the foot on lateral foot radiograph.
Calcaneal Inclination Angle | Initial evaluation of the participant
  Angle formed by a line tangent to the inferior cortex of the calcaneus and an horizontal reference line of the plantar plane on lateral foot radiograph.
Lateral Talo-first metatarsal Angle | Initial evaluation of the participant
  Angle formed by the longitudinal axis of the first metatarsal shaft and the longitudinal axis of the talus on lateral foot radiograph.

SECONDARY OUTCOMES:
Popliteal angle | Initial evaluation of the participant
  Popliteal angle was defined as the acute angle between tibia and femur when the knee joint was passively extended with the hip flexed 90 degrees.
Ankle range of motion | Initial evaluation of the participant
  The degree of flexion, extension, inversion, and eversion of the ankle joint that measured regarding the neutral zero methods.
The degree of spasticity of the certain muscles of the lower extremities | Initial evaluation of the participant
  The tonus of hip flexor, hip adductor, knee extensor, knee flexor, ankle plantar flexor, and ankle invertor muscles will be evaluated by the Modified Ashworth Scale. Achilles' tendon tightness will be evaluated by the Silfverskiöld Test.

OTHER OUTCOMES:
Gait pattern | Initial evaluation of the participant
  Based on the visual evaluation, the patient's gait pattern will be determined. (true crop, visible crop, squat gait, knee jump or mixed)

CONTACTS AND LOCATIONS:
Overall Officials: Murat Zinnuroğlu, MD, Principal Investigator — Gazi University Faculty of Medicine; Levent Karataş, MD, Principal Investigator — Gazi University Faculty of Medicine
Locations (1):
- Gazi University Hospital, Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Min JJ, Kwon SS, Sung KH, Lee KM, Chung CY, Park MS. Progression of planovalgus deformity in patients with cerebral palsy. BMC Musculoskelet Disord. 2020 Mar 3;21(1):141. doi: 10.1186/s12891-020-3149-0. PMID 32127007
- [Background] Butler RJ, Hillstrom H, Song J, Richards CJ, Davis IS. Arch height index measurement system: establishment of reliability and normative values. J Am Podiatr Med Assoc. 2008 Mar-Apr;98(2):102-6. doi: 10.7547/0980102. PMID 18347117
- [Background] Drefus LC, Kedem P, Mangan SM, Scher DM, Hillstrom HJ. Reliability of the Arch Height Index as a Measure of Foot Structure in Children. Pediatr Phys Ther. 2017 Jan;29(1):83-88. doi: 10.1097/PEP.0000000000000337. PMID 27984478